CLINICAL TRIAL: NCT06454149
Title: Establishment of a Cohort for Investigating the Pathophysiology of Gastric MALT Lymphoma
Brief Title: Cohort Study for Gastric MALT Lymphoma
Acronym: HUG-MALToma
Status: Recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: Kangbuk Samsung Hospital (Other); Korea University Ansan Hospital (Other)
Responsible Party: Principal Investigator, Cheol Min Shin, Professor, Seoul National University Hospital
Other Study IDs: HUG-MALToma
Record Dates: First submitted 2024-06-06; First posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Gastric MALT Lymphoma
MeSH Terms: interventions — MALT1 protein, human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MALT lymphoma: Patients who were newly diagnosed as gastric MALT lymphoma
  Interventions: Other: MALT lymphoma
- Control group: Patients who underwent
  1. diagnosed upper endoscopy for dyspepsia and had chronic gastritis,
  2. therapeutic upper endoscopy for gastric hyperplastic polyps, or
  3. screening upper endoscopy without any symptoms.

INTERVENTIONS:
Other: MALT lymphoma — New diagnosis with gastric MALT lymphoma
  Groups: MALT lymphoma

SUMMARY:
The goal of this observational study is to establish clinical data and tissue repository in patients with gastric MALT lymphoma and controls.

Participants will be asked to provide clinical information and various tissues (saliva, gastric mucosa, and feces).

ELIGIBILITY:
Inclusion Criteria:

[MALT lymphoma group]

* Newly diagnosed as gastric MALT lymphoma [Control group]
* Patients who underwent

  1. diagnosed upper endoscopy for dyspepsia and had chronic gastritis,
  2. therapeutic upper endoscopy for gastric hyperplastic polyps, or
  3. screening upper endoscopy without any symptoms.

Exclusion Criteria:

* History of gastric or other malignancy
* Use of antibiotics or probiotics within 4 weeks
* Uncontrolled chronic illnesses

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Eligible patients who visited participating hospital will be asked, and upon providing informed consent, will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-06-06 (Actual); Primary Completion 2028-06-05 (Estimated); Study Completion 2031-06-05 (Estimated)

PRIMARY OUTCOMES:
Remission of gastric MALT lymphoma | Within 3 years from diagnosis
  Remission of gastric MALT lymphoma

SECONDARY OUTCOMES:
Eradication of H. pylori infection | Within 6 month from eradication therapy
  Eradication of H. pylori infection

CONTACTS AND LOCATIONS:
Locations (3):
- South Korea (3):
  - Korea University Ansan Hospital, Ansan-si, Gyeonggi-do
  - Cheol Min Shin, Seongnam-si, Gyeonggi-do
  - Kangbuk Samsung Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to data protection policy of the participating institutions.

REFERENCES:
- [Background] Zucca E, Arcaini L, Buske C, Johnson PW, Ponzoni M, Raderer M, Ricardi U, Salar A, Stamatopoulos K, Thieblemont C, Wotherspoon A, Ladetto M; ESMO Guidelines Committee. Electronic address: clinicalguidelines@esmo.org. Marginal zone lymphomas: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2020 Jan;31(1):17-29. doi: 10.1016/j.annonc.2019.10.010. Epub 2019 Dec 4. No abstract available. PMID 31912792
- [Background] Di Rocco A, Petrucci L, Assanto GM, Martelli M, Pulsoni A. Extranodal Marginal Zone Lymphoma: Pathogenesis, Diagnosis and Treatment. Cancers (Basel). 2022 Mar 29;14(7):1742. doi: 10.3390/cancers14071742. PMID 35406516
- [Background] Tanaka T, Matsuno Y, Torisu T, Shibata H, Hirano A, Umeno J, Kawasaki K, Fujioka S, Fuyuno Y, Moriyama T, Esaki M, Kitazono T. Gastric microbiota in patients with Helicobacter pylori-negative gastric MALT lymphoma. Medicine (Baltimore). 2021 Sep 24;100(38):e27287. doi: 10.1097/MD.0000000000027287. PMID 34559138
- [Background] Lemos FFB, Silva Luz M, Rocha Pinheiro SL, Teixeira KN, Freire de Melo F. Role of non-Helicobacter pylori gastric Helicobacters in helicobacter pylori-negative gastric mucosa-associated lymphoid tissue lymphoma. World J Gastroenterol. 2023 Aug 28;29(32):4851-4859. doi: 10.3748/wjg.v29.i32.4851. PMID 37701138